CLINICAL TRIAL: NCT03084159
Title: Multi-disciplinary Participatory Design of a Process to Deliver a CKD Diagnosis in Primary Care
Acronym: EPIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Julie Wright-Nunes, Associate Professor, University of Michigan
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: HUM00118819; 4K23DK097183-04 (NIH)
Record Dates: First submitted 2017-02-20; First posted 2017-03-20 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Participatory design and intervention (Experimental): Patients in this arm will receive the intervention of using an education worksheet during their appointment with their provider. They will be asked to complete post intervention surveys (for feasibility and feedback prior to actual trial enrollment). Providers and staff at this site have been involved in the design of the intervention process, to make it streamlined and efficient for application in practice.
  Interventions: Behavioral: Education worksheet
- Intervention Only (Experimental): This arm include new patients at the initial site that also received the intervention of using an education worksheet during their appointment and filled out post intervention surveys. Some of these providers/staff were not involved in the initial design of the intervention.
  Interventions: Behavioral: Education worksheet
- Usual Care (No Intervention): A second site included usual care, which did not include the intervention. Participants were given post visit surveys similar to those in the two other study / intervention arms. This site served as a usual care comparison.

INTERVENTIONS:
Behavioral: Education worksheet — Patients who screen positive for CKD and give written informed consent to be a part of the study will have their chart flagged for the medical assistant and provider to give the education worksheet intervention. The education worksheet has been developed to be used as an electronic tool within the Electronic Medical Record. The provider will review it with the patient during the visit. A paper copy will print out for the patient at the end of the visit.
  Other Names: Education Activation Worksheet
  Arms: Intervention Only; Participatory design and intervention

SUMMARY:
This study will use an adapted education worksheet to support patient-centered chronic kidney disease (CKD) communication, shared decision making, and patient engagement and will test its impact on intermediate patient modifiable characteristics in a primary care practice with patients who have pre-dialysis CKD.

The study team will enroll up to 100 patients with chronic kidney disease (CKD) from a primary care clinic to start. Patients will receive the intervention, which consists of the physicians using the education worksheet during appointments with patients, and patients and providers will complete surveys about its use and to measure impact on knowledge and other areas related to patient outcomes.

Once initial user testing is complete, the study team plans to submit an amendment to expand on this trial and incorporate comparison sites. This will be submitted and receive IRB approval prior to participant involvement.

The study hypothesis is that patients who receive the intervention will have greater knowledge about their CKD diagnosis, higher satisfaction with provider communication, and higher scores related to managing CKD to keep themselves healthy compared to control populations.

DETAILED DESCRIPTION:
Amendment on 12/2018: The enrollment numbers were updated to include the control group.

Clarification 9/2021: After initial feasibility was assessed, the initial site was used additionally to enroll for the "second arm", rather than a new site as originally intended. A second site was then used for the control population.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Have an estimated glomerular filtration rate (eGFR) of less than 60 ml/min/1.73 m2
* Able to read and understand English without an interpreter
* Diagnosed with chronic kidney disease on record

Exclusion Criteria:

* Patients with renal transplant or on dialysis
* Patients who have documented or provider known cognitive impairment or vision impairment that will prohibit meaningful interaction with education activation worksheet
* Patients who are not aware of their CKD diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
Level of objective understanding of CKD as measured by the Kidney Knowledge Survey (KiKS) | Length of doctor's appointment, e.g., 1-2 hours
  This will measure objective kidney disease knowledge, based on a score of 0-100, where 0 means poor level of kidney knowledge, and 100 means good level of kidney knowledge. The KiKS was developed by Dr. Wright.
Level of perceived understanding of CKD as measured by the Perceived Kidney Knowledge Survey (PiKS) | Length of doctor's appointment, e.g., 1-2 hours
  This will measure subjective kidney knowledge. Score range is 1-4, where 1 is low level of perceived kidney knowledge, and 4 is high level of perceived kidney knowledge. The PiKS was developed by Dr. Wright.

SECONDARY OUTCOMES:
Level of positive perception of patient-provider communication as measured by the Patient Communication Assessment Tool (CAT) | Length of doctor's appointment, e.g., 1-2 hours
  This assesses the quality of physician to patient and physician's staff to patient communication. Score range is 1-5, where 1 means negative perception of communication and 5 means positive perception of communication.
Level of mental anxiety/stress related to condition as measured by the adapted NDBCSS scale | Length of doctor's appointment, e.g., 1-2 hours
  The 19-item NDBCSS (Newly Diagnosed Breast Cancer Stress Scale) is adapted to form the 21-item scale in the patient survey to measure stress associated with CKD. The score range is 1-4, where 1 means high level of stress associated with CKD and 4 means low level of stress associated with CKD.
Level of energy/fatigue and emotional well-being as measured by the SF-36 mental health component | 4 weeks
  The SF-36 mental health component is a 9-item scale that measures energy/fatigue and emotional well-being in the past 4 weeks.Score range is 0-100, where 0 means poor emotional well-being and low energy and 100 means good emotional well-being and high energy.

OTHER OUTCOMES:
Level of positive assessment of care as measured by the Patient Assessment of Care for Chronic Conditions (PACIC) scale | 6 months
  This is a 11-item scale evaluating patient assessment of the quality of care that patients received in the past 6 months. Score range is 1-5, where 1 means poor assessment of quality of care and 5 means good assessment of quality of care.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Wright-Nunes, MD, MPH, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Canton Health Center, Canton, Michigan
  - Northville Health Center, Northville, Michigan

IPD SHARING:
Plan to Share IPD: No